CLINICAL TRIAL: NCT06613581
Title: Patient-empowered Remote Oncology: the Prospective, Multicentre Implementation Study - the PROMISE
Brief Title: Patient-led Follow-up from Home After Surgery for Colorectal Carcinoma
Acronym: PROMISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Lifesignals Inc. (Unknown); YourBio Health (Unknown); TU Delft (Unknown); Amphia Hospital (Other); Leiden University Medical Center (LUMC) (Unknown); Franciscus Gasthuis & Vlietland (location Rotterdam) (Unknown)
Responsible Party: Principal Investigator, D.J. (Dirk) Grünhagen, Surgical oncologist, MD, PhD, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NL84788.078.23; 84788 (Other: ToetsingOnline (ABR-form))
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Carcinoma (CRC)
Keywords: Colorectal carcinoma; Home-based follow-up; Patient-led; Capillary blood sampling; Biosensor; EORTC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients included in the study will be followed-up according to the home-based follow-up protocol. The PROMISE study is an implementation study, to further develop and improve home-based follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implementation of home-based follow-up (Experimental): All patients within the PROMISE study are included in the 'experimental' arm. The study is set up as an implementation study, meaning that the home-based method of follow-up is applied to all patients in the study.
  Interventions: Other: Home-based follow-up

INTERVENTIONS:
Other: Home-based follow-up — Follow-up after surgery for colorectal carcinoma, performed from home, within the bounds of the Dutch National guidelines

SUMMARY:
The primary goal of the patient-led follow-up from home, is the improvement of quality of life and the reduction of stress in patients, while obtaining a more complete picture of their health status.

A series of assessments are performed in the home setting:

* Blood withdrawal for CEA determination
* Quality of life questionnaires to assess both mental and physical symptoms
* Vital parameters using a Smart Sensor

DETAILED DESCRIPTION:
Primary Objective: To further develop and evaluate a personalised patient-centred surveillance programme including a feedback platform for patients after curative treatment for CRC in terms of health-related quality of life (HRQoL) and significantly decrease the number of in-hospital appointments, by relocating the follow-up care to the home-setting. The goal is for this surveillance program to be non-inferior to standard of care follow-up at 36 months, in terms of quality of life. The quality of life in patients will be assessed with the EQ 5D-5L questionnaire and compared to median EQ-5D-5L scores for patients receiving standard of care follow-up. In current literature, the median HRQoL VAS score for patients after surgery for CRC is 62.05 points (1).

The second goal of the program is to relocate part of the in-hospital follow-up care to the home-setting. In standard of care follow-up, at 36 months patients would have had 10 in-hospital appointments. The effect of the PROMISE study on the number of in-hospital appointments, will be assessed at 36 months postoperatively.

The PROMISE study is a multi-centre prospective regional implementation study of a personalised patient-centred surveillance program including a feedback platform for patients after curative treatment for CRC.

All patients who underwent surgery with curative intent for non-metastatic CRC with scheduled postoperative surveillance are potentially eligible.

Follow-up in this study is performed according to the acting Dutch national guidelines. Current guidelines advocate CEA level measurements to be performed every 3-6 months for first 2 years after surgery and every 6-12 months for years 3 to 5. Medical imaging (thoracic and abdominal CT) should be performed 1 year postoperatively. Changes to the Dutch national guidelines during the course of the study will be implemented accordingly into the follow-up.

Within this study surveillance will for the greater part be performed at home:

* Serum CEA level monitoring is performed using the automatic capillary blood withdrawal device (TAP-II) - every 6 months during the first two years and every 12 months thereafter
* Vital parameters will be measured with a LifeSignals Multi-parameter Remote Monitoring System - every 3 months during the first two years and every 6 months thereafter
* QoL is measured with the use of questionnaires - every 3 months during the first two years and every 6 months thereafter
* One scheduled in hospital evaluation with medical imaging (according to national guidelines) performed 1 year after surgical treatment

ELIGIBILITY:
inclusion criteria

* Age ≥ 21 years
* Histologically confirmed colorectal adenocarcinoma without distant metastasis and treated with curative intent surgical resection less than 6 months ago
* Scheduled or currently undergoing postoperative surveillance according to national guidelines
* Written informed consent by the patient
* Access to a smartphone

Exclusion criteria

* Patients with a severely complicated postoperative course, needing in hospital follow- up longer than 6 months postoperatively
* Patients enrolled in other studies that require strict adherence to any specific follow-up practice with regular imaging - yearly or more frequent - of the abdomen and/or thorax
* Patients with comorbidity or other malignancy that requires imaging of the abdomen and/or thorax every year or more frequent
* Patients with active implantable devices - e.g. pacemaker or implantable defibrillator
* Inability to complete the questionnaires due to illiteracy and/or insufficient proficiency of the Dutch language

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 36 months
  The primary outcome of this study is to evaluate non-inferiority of the study follow-up with respect to the EQ-5D-5L score at 36 months of follow-up, which starts within 6 months of resection of the primary tumour.
Number of in hospital visits | 36 months
  The second primary outcome consists of significantly decreasing the number of in-hospital appointments, by relocating this follow-up care to the home setting. This will be assessed at 36 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J. Grunhagen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (5):
- Netherlands (5):
  - Amphia Hospital, Breda, North Brabant
  - IJsselland Hospital, Capelle aan den IJssel, South Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Franciscus Gasthuis and Vlietland, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No
IPD can be shared, but exclusively upon reasonable request with the affiliated researchers